CLINICAL TRIAL: NCT04030845
Title: Chinese Multicenter Prospective Registry of Breast Cancer Patient Reported Outcome -Reconstruction and Oncoplastic Cohort
Brief Title: Patient Report Outcome-Reconstruction and Oncoplastic Cohort
Acronym: PRO-ROC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); First Hospital of China Medical University (Other); Guangdong Provincial People's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The First Affiliated Hospital of Air Force Medicial University (Other); Hunan Province Cancer Hospital and the Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University (Unknown); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); First Affiliated Hospital of Zhejiang University (Other); The First Affiliated Hospital of Xiamen University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Hubei Cancer Hospital (Other); The Affiliated Hospital of Qingdao University (Other); First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jiong Wu, Professor, Department of Breast Surgery Vice President Cancer Hospital/Institute, Fudan University, Fudan University
Other Study IDs: SCHBCC-N023
Record Dates: First submitted 2019-07-12; First posted 2019-07-24 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Patient Reported Outcome Measures; Breast Reconstruction; Oncoplastic Breast-conserving Surgery; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammaplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- breast reconstruction
  Interventions: Procedure: breast reconstruction
- oncoplastic breast-conserving surgery
  Interventions: Procedure: oncoplastic breast-conserving surgery

INTERVENTIONS:
Procedure: breast reconstruction — The breast reconstruction mainly included autologous tissue flaps (latissimus dorsi myocutaneous flaps, pedicled tansverse rectus abdominis myocutaneous flaps, free transverse rectus abdominis musculocutaneous flaps, deep inferior epigastric artery perforator flaps, etc.), implant based breast reconstruction, autologous flaps combined with implant reconstruction, fat graft, etc.
  Groups: breast reconstruction
Procedure: oncoplastic breast-conserving surgery — The oncoplastic breast-conserving surgery were mainly those surgeries using volume displacement or volume replacement techniques.
  Groups: oncoplastic breast-conserving surgery

SUMMARY:
Available studies that focused on patient-reported outcomes (PROs) were mainly from one institution or of small sample size. The variations across hospitals and regions were not fully analyzed. A multicenter prospective patient report outcome-reconstruction and oncoplastic cohort (PRO-ROC) will be planned to assess the PROs for Chinese breast cancer patients who will undergo breast reconstruction or oncoplastic breast-conserving surgery (OBCS). The inclusion criteria are female breast cancer patients >18 years old, who will undergo breast reconstruction (BR) or OBCS. This cohort will include at least 10000 patients (about 5000 patients who undergo BR, and 5000 patients who undergo OBCS). The exposures were the surgery types: BR and OBCS regardless of the techniques and materials they used. The primary endpoint will be PROs, which include BREAST-Q, quality of life (EORTC QLQ-C30), EORTC QLQ-BR23). This study follows the Helsinki Declaration and Chinese rules. All patients will be asked to to sign the informed consent and will be followed up 24 months after operations. All data will be collected using an app software.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer patients;
2. Adult (>18 years old);
3. Female;
4. Must undergo breast reconstruction or oncoplastic breast-conserving surgery;

Exclusion Criteria:

1. Younger (<18 years old);
2. Male;
3. Stage IV breast cancer patients;
4. Refuse to undergo breast reconstruction or oncoplastic breast-conserving surgery.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients are confirmed by histopathologic evaluation without distant metastasis (M0). The patients must fulfill indications of breast cancer surgery according to NCCN clinical guidelines, and do not have any absolute contraindications.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in BREAST-Q score | Change from baseline at 1 year and 2 years post-operatively.
  The Breast-Q© is a patient reported outcome measure (PROM) for breast surgery that was rigorously developed to accurately measure patient reported satisfaction and quality of life (QOL). (http://www.mskcc.org/mskcc/shared/Breast-Q/index.html). The BREAST-Q was developed and validated with adherence to international guidelines. This PROM is composed of six scales that address: 1) psychosocial well-being, 2) physical well-being, 3) sexual well-being, 4) satisfaction with breasts, 5) satisfaction with outcome, and 6) satisfaction with care. Each module generates a Q-score on a 0-100 scale that can be used for quantitative analysis to enable statistical comparison of the pre- to the post-operative state.
Change from baseline in health-related quality of life measured by EORTC QLQ-C30 | Change from baseline at 1 year and 2 years post-operatively.
  To compare change in Quality of Life, as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30 (Version 3)) from baseline at 1 year and 2 years post-operatively. The EORTC QLQ-C30 (Version 3) uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome. The EORTC QLQ-C30 (Version 3) uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Change from baseline in health-related quality of life measured by EORTC QLQ-BR23 | Change from baseline at 1 year and 2 years post-operatively.
  EORTC QLQ-BR-23 consists of 23 questions related to breast cancer. The questionnaire will be self-administered and will be given in patient's mother tongue. EORTC-QLQ-BR23: included functional scales (body image, sexual functioning, sexual enjoyment, and future perspective) and single item symptoms scales (systemic therapy side effects, breast symptoms, arm symptoms, and upset by hair loss). Questions used 4-point Likert scale (1 'Not at All' to 4 'Very Much'). Scores averaged and transformed to 0-100 scale. High score for functional scale=high/healthy level of functioning. High score for single item=high level of symptomatology/problems.

SECONDARY OUTCOMES:
Rates of complications | up to 24 months
  complications includes overall complication，implant loss, seroma, wound-skin infection, nipple or skin flap necrosis, hematoma, reoperation, wound dehiscence, capsular contracture
Change from baseline in cosmetic scores rated by patients | Change from baseline at 1 year and 2 years post-operatively.
  Cosmetic outcomes scored by the patients. Cosmetic scores rates from 0 to 5, which 0 means very dissatisfied, and 5 means very satisfied.
breast aesthetics | up to 24 months
  An anterior view picture of the patient will be taken with the patients hands on the hips at baseline (before surgery), postoperative 3, 12 and 24 months in order to assess breast aesthetics. A panel of at least three independent observers blinded to patient identity, treatment allocation, and radiotherapy center scored the photographs. Breast size and surgical deficit were scored from the baseline photographs on a 3-point scale (small, medium, large). After radiotherapy, breast appearance change (none/mild/marked) was scored on a pair of photographs with standard positions in comparison with the baseline photograph.
Overall survival | up to 24 months
  Overall survival (OS) was defined as the time from beginning treatment to the time of death from any cause or the date of last contact if death was not recorded before the cutoff date.
Recurrence-free survival | up to 24 months
  Recurrence-free survival (RFS) was calculated as time from breast cancer diagnosis until locoregional (LRRFS) or distant recurrence (DRFS) or death due to breast cancer, whichever came first.

OTHER OUTCOMES:
change from baseline in Visual Analog Score for pain | Change from baseline at 1 day, 3 days, 7 days, 3 months, 1 year and 2 years post-operatively.
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. Pain will be evaluated according to the Visual-analogue scale (VAS) varying from 0 to 10 with a higher score indicating a higher level of pain where 0 represents no pain and 10 represents the strongest pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer Center, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Chi W, Zhang Q, Li L, Chen M, Xiu B, Yang B, Wu J. Immediate Breast Reconstruction After Neoadjuvant Chemotherapy: Factors Associated With Surgical Selection and Complications. Ann Plast Surg. 2023 Jul 1;91(1):48-54. doi: 10.1097/SAP.0000000000003574. Epub 2023 May 19. PMID 37216212
- [Derived] Li L, Yang B, Li H, Yin J, Jin F, Han S, Liao N, Shi J, Ling R, Li Z, Ouyang L, Wang X, Fu P, Ouyang Z, Ma B, Wu X, Wang H, Liu J, Shao Z, Wu J. Chinese multicentre prospective registry of breast cancer patient-reported outcome-reconstruction and oncoplastic cohort (PRO-ROC): a study protocol. BMJ Open. 2019 Dec 15;9(12):e032945. doi: 10.1136/bmjopen-2019-032945. PMID 31843846